CLINICAL TRIAL: NCT01085019
Title: Investigation of the Impact of Spices and Herbs on Endothelial Function and Other CVD Risk Factors in Men and Women.
Brief Title: Impact of Spices and Herbs on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: McCormick Canada Co (Unknown)
Responsible Party: Principal Investigator, Charles Couillard, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INAF-2009-253
Record Dates: First submitted 2010-03-09; First posted 2010-03-11 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Endothelial Function
Keywords: Endothelial function; Cardiovascular risk factors; Spices; Herbs; Antioxidant
MeSH Terms: interventions — ginger extract; black pepper oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dietary supplement: Cinnamon (Experimental)
  Interventions: Dietary Supplement: Cinnamon
- Dietary supplement: Oregano (Experimental)
  Interventions: Dietary Supplement: Oregano
- Dietary supplement: Ginger (Experimental)
  Interventions: Dietary Supplement: Ginger
- Dietary supplement: Rosemary (Experimental)
  Interventions: Dietary Supplement: Rosemary
- Dietary supplement: Black pepper (Experimental)
  Interventions: Dietary Supplement: Black pepper
- Dietary supplement: Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cinnamon — 2.8g/day of cinnamon in capsules during 4 weeks.
  Arms: Dietary supplement: Cinnamon
Dietary Supplement: Oregano — 2.8g/day of oregano in capsules during 4 weeks.
  Arms: Dietary supplement: Oregano
Dietary Supplement: Ginger — 2.8g/day of ginger in capsules during 4 weeks.
  Arms: Dietary supplement: Ginger
Dietary Supplement: Rosemary — 2.8g/day of rosemary in capsules during 4 weeks.
  Arms: Dietary supplement: Rosemary
Dietary Supplement: Black pepper — 2.8g/day of black pepper in capsules for 4 weeks.
  Arms: Dietary supplement: Black pepper
Dietary Supplement: Placebo — 2.8 g/day of placebo in capsules (corn starch) during 4 weeks.
  Arms: Dietary supplement: Placebo

SUMMARY:
The general objective of the study is to investigate the effects of the daily consumption of spices and herbs for four (4) consecutive weeks in endothelial function and cardiovascular risk factors of men and postmenopausal women.

DETAILED DESCRIPTION:
The purpose is to assess whether the polyphenol/antioxidant content of different spices will affect endothelial function and other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 yrs
* Men and postmenopausal women
* Waist girth >102cm (men) or >88cm (women)
* LDL-C > 2.8 mmol/L
* Framingham 10-yr risk score < 10%
* Marginal endothelial dysfunction
* Non smoker

Exclusion Criteria:

* Medication for lipid, hypertension, diabetes
* History of CVD, diabetes, other endocrines disorders
* Pre-menopausal women
* Alcohol consumption > 1 drink per day
* Unusual dietary habits (e.g. vegetarism)
* Chronic use of supplements (estrogens, vitamins, minerals or flavonoids)
* Aversion or intolerance for spices and/or herbs
* Injury to fingers or amrs that would interfere with endothelial function measurement

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function measured by endopat system (the endothelium-mediated changes in vacular tone) | at week 0 and week 4

SECONDARY OUTCOMES:
Circulating level of plasma lipoproteins-lipids | at week 0 and week 4
Oxidative stress | at week 0 and week 4
Endothelial activation and inflammatory markers | at week 0 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Charles Couillard, Ph.D, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - Richardson Centre of Functional Foods and Nutracuticals, Winnipeg, Manitoba
  - Institute of Nutraceuticals and Functional Foods, Québec, Quebec

REFERENCES:
- [Derived] Carnovale V, Paradis ME, Gigleux I, Ramprasath VR, Couture P, Jones PJ, Lamarche B, Couillard C. Correlates of reactive hyperemic index in men and postmenopausal women. Vasc Med. 2013 Dec;18(6):340-6. doi: 10.1177/1358863X13507975. PMID 24292639